CLINICAL TRIAL: NCT04226846
Title: A Clinical Feasibility Study of the Bios Device for Continuous Glucose Monitoring in Subjects With Type 1 or Type 2 Diabetes Mellitus
Brief Title: Feasibility Trial of the Bios Device for Continuous Glucose Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GraphWear Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GRAPHWEAR 001
Record Dates: First submitted 2019-12-30; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is an open-label, prospective, within-subject comparison of the Bios device readings versus venous blood sample glucose readings, glucose readings from a Dexcom CGM and an SMBG device in subjects previously diagnosed with Type 1 or Type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age;
2. Subject has had a diagnosis of diabetes mellitus either Type I or Type II;
3. For insulin-using subjects only: subject will not inject insulin or wear an insulin pump insertion set within a 10 cm distance of any Bios device;
4. Subject able to wear multiple CGM devices simultaneously;
5. Subject is either a patient diagnosed with Type I diabetes mellitus currently wearing a Dexcom CGM device or a patient diagnosed with Type II diabetes mellitus who will agree to use a Dexcom CGM device during participation in the study. There are no restrictions on the model of the Dexcom CGM device.
6. Subject agrees to provide a log of medications (prescription and over-the-counter) and dietary supplements (e.g., vitamins) taken during the study period, including dosage;
7. Subject has a smart device that complies with the requirements listed in Attachment 1 of this protocol and is willing to download and run the GraphWear Patient application on their device;
8. Subject is able to read and understand the Informed Consent Form and has voluntarily provided written informed consent;
9. In the Principal Investigator's opinion, subject is able to be compliant with provisions laid out in this protocol.

Exclusion Criteria:

1. Subjects with any physical or behavioral disorder, which, in the opinion of the Principal Investigator, may interfere with the use of the device or compliance with the study protocol;
2. Subject has any of the following:

   * a skin condition that precludes wearing of the device;
   * a known allergy that precludes wearing of the device;
   * tattoos or other skin alterations that may interfere with device placement and/or operation;
3. History of substance abuse within 6 months of study start;
4. Use of any illicit drugs during the duration of the study period;
5. Marijuana use during the duration of the study period;
6. If female, subject is pregnant or nursing;
7. Subject is on active dialysis;
8. Subjects whom the Principal Investigator believes may not be an appropriate candidate for this device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously diagnosed with Type 1 or Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Comparison between Bios device readings and glucose values | 2 weeks
  The primary objective of this study is to compare the glucose measurements collected by the Bios device to glucose values measured with a blood glucose lab analyzer (e.g., YSI), glucose values obtained with a self-monitoring blood glucose device (SMBG) and readings from the Dexcom System in subjects previously diagnosed with Type 1 or Type 2 diabetes mellitus.

CONTACTS AND LOCATIONS:
Locations (1):
- Diablo Clinical Research, Inc, Walnut Creek, California, United States